CLINICAL TRIAL: NCT03846492
Title: Targeting Brain Physiology to Treat Neuropsychiatric Symptoms of Dementia Using TMS-EEG and tDCS
Acronym: tTED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: BrightFocus Foundation (Other)
Responsible Party: Principal Investigator, Sanjeev Kumar, Staff Psychiatrist and Clinician Scientist, Medical Head of Geriatric Clinical Research, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 093/2018
Record Dates: First submitted 2019-02-08; First posted 2019-02-19 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Alzheimer Disease; Dementia, Mixed; Dementia; Behavior Problem; Dementia, Alzheimer Type
Keywords: Dementia; Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation; tDCS; TMS; TMS-EEG; MRI; Agitation; Alzheimer's disease; Neuropsychiatric symptoms; Agitation in dementia; Mixed dementia; Non-invasive brain stimulation
MeSH Terms: conditions — Alzheimer Disease; Mixed Dementias; Dementia; Mental Disorders; Psychomotor Agitation; Aberrant Motor Behavior in Dementia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Individuals with AD + agitation will receive a 2 week course of active/sham cathodal tDCS to frontal brain region in a double blind 1:1 randomized control design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS (Experimental): The direct current will be delivered at 2 mA intensity via rubber electrodes in saline- soaked sponges for 30 min per day for 2 weeks, 5 days/week. Inhibitory stimulation will be delivered to the frontal lobes.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- sham tDCS (Sham Comparator): Sham tDCS will use the same parameters except that the device will automatically turn off after a certain duration.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS is a non-invasive brain stimulation modality that does not require general anesthesia or surgical implantation of a device. tDCS utilizes low intensity electrical current either to increase cortical excitability with an anodal electrode or to suppress cortical excitability with a cathodal electrode. It uses 3 AAA batteries to deliver direct current via rubber electrodes enclosed in saline soaked sponges.

SUMMARY:
Agitation and aggression impose a tremendous burden on the individuals living with dementia, their families, caregivers, and healthcare systems. Neuropsychiatric symptoms of dementia (NPS) affect up to 80% of patients with Alzheimer's dementia (AD). The mechanisms of agitation in AD are poorly understood and the current interventions are only modestly effective while having serious adverse effects. In this study, the investigators propose to assess the mechanisms and treatment of neuropsychiatric symptoms in AD with the use of non-invasive, brain stimulation approaches. By applying magnetic stimulation to the surface of the head (transcranial magnetic stimulation - TMS) combined with electroencephalography (EEG), the investigators will be able to study the mechanisms of agitation and advance our understanding of AD. Further, the investigators will evaluate if transcranial direct current stimulation (tDCS) is effective to treat agitation dementia.

DETAILED DESCRIPTION:
Alzheimer's dementia (AD) and related neurodegenerative diseases are inflicting a global healthcare crisis. Neuropsychiatric symptoms including agitation and aggression affect up to 80% of patients with AD. Among these symptoms, agitation and aggression are the most burdensome for patients, families, caregivers, and the health care system. The mechanisms of agitation in AD are poorly understood and the current interventions are only modestly effective while having serious adverse effects.

In this study, the investigators propose to assess the mechanisms and treatment of neuropsychiatric symptoms in AD with the use of non-invasive, brain stimulation approaches. Agitation/aggression is associated with abnormalities in the balance of cortical excitation/inhibition. Transcranial magnetic stimulation (TMS) using single and paired pulse TMS paradigms such as long interval cortical inhibition (LICI) and short interval intracortical inhibition (SICI) can assess this cortical excitation/inhibition balance in vivo. The investigators will use TMS, combined with electroencephalography (EEG), to assess cortical excitation/inhibition balance in the dorsolateral prefrontal cortex (DLPFC) of participants with AD with and without agitation/aggression and age matched healthy comparators.

Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that uses a very low intensity electric current to modulate cortical excitability and brain plasticity. tDCS can restore excitation and inhibition balance by altering GABA and glutamate activity in the brain. tDCS can be safely administered to awake persons and is very well tolerated. Studies in healthy individuals and patients with AD have shown that tDCS applied to frontal brain regions can enhance cognitive function. Further, tDCS applied to frontal brain regions can improve depressive symptoms. The effects of tDCS on neuropsychiatric symptoms are not known. In this study, the investigators will use tDCS applied to the frontal brain regions to target deficits in inhibition and symptoms of agitation/aggression in AD.

This study will be done over a period of 3 years at Centre for Addiction and Mental Health Geriatric Psychiatry Division and Temerty Centre for Therapeutic Brain Intervention. The investigators will recruit and enroll 30 individuals with AD + Agitation (mild to moderate agitation), 30 individuals with AD without agitation and 30 older healthy individuals. Medical work up will be done as part of clinical care prior to study enrollment to rule out medical causes of agitation. Clinical and cognitive assessments will be performed to characterize participants at baseline. The investigators will assess cortical inhibition using TMS EEG at baseline in the three groups. Individuals with AD + agitation will then receive a 2 week course of active/sham cathodal tDCS to frontal brain region in a double blind 1:1 randomized control design. Assessment of cortical inhibition using measures identical to baseline will be done at the end of tDCS course. The investigators will also repeat clinical and cognitive assessments after tDCS course and 2 weeks later. Measures of cortical inhibition will first be compared between HC and AD, and between AD and AD + Agitation groups. The treatment effects on clinical symptoms, cortical inhibition and the rate adverse events will be compared between active and sham tDCS groups.

During the Covid-19 pandemic, the study has been modified to be administered in a hybrid manner to accommodate both in-person and virtual assessments. Clinical and cognitive assessments can be done in-person or remotely. The initial tDCS course will be conducted in-person with the research staff. The remaining tDCS intervention will be completed onsite or at the participant's home with virtual supervision from the research team.

ELIGIBILITY:
Participants with AD+Agitation

Inclusion:

1. Age 50 years or older.
2. Participant or substitute decision maker able and willing to provide informed consent.
3. Dementia due to probable or possible AD as defined by NIA-AA criteria.
4. Presence of mild to moderate agitation and/or aggression as defined by: Agitation in cognitive disorders. International Psychogeriatric Association Provisional Consensus Clinical and Research Definition.
5. Availability of a support person to accompany the participant to study appointments and provide collateral information as needed.
6. If taking medication for neuropsychiatric symptoms, the dose should be stable for at least 1 week.

Exclusion:

1. Psychiatric diagnosis other than dementia significantly impacting the presentation.
2. Presence of delirium or other acute medical condition significantly contributing to agitation/aggression or making the study participation unsafe for a participant.
3. Any contraindication to TMS or tDCS.
4. Any other condition that in the opinion of principal investigator will make the study participation unsafe or non-feasible for the participant.
5. Currently taking anticonvulsants or benzodiazepines at a dose sufficient to cause interference with TMS-EEG.

Participants with AD without aggression

All the above inclusion/exclusion criteria except meeting the inclusion criterion 4 pertaining to agitation/aggression. Participants with significant agitation/aggression will be excluded from this group.

Healthy comparator participants

Inclusion:

1. Age 50 years or older.
2. Able and willing to provide informed consent.
3. Free from any significant neurological disorder.

Exclusion:

1. Lifetime DSM-5 diagnosis other than simple phobias or adjustment disorder.
2. Any Contraindication to TMS.
3. Currently taking anticonvulsants or benzodiazepines at a dose sufficient to cause interference with TMS-EEG.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-04-24 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Long Interval Cortical Inhibition (LICI), a TMS paradigm, will be used to assess the extent of cortical inhibition | Baseline
  LICI will be measured using single and paired TMS pulses applied to the Dorsolateral Prefrontal Cortex (DLPFC). LICI will be compared between the 3 groups (AD, AD+agitation and healthy comparators).

SECONDARY OUTCOMES:
Short Interval Cortical Inhibition (SICI), another TMS paradigm, will be used to assess the extent of cortical inhibition | Baseline
  SICI will be measured using single and paired TMS pulses applied to the DLPFC and motor cortex. SICI will be compared between the 3 groups (AD, AD+agitation and healthy comparators).
The rate of successful completion of the 2 week tDCS treatment course | Approximately 2 weeks after baseline
  This will be assessed by the successful completion of the intervention in at least 80% of participants without any treatment associated serious adverse effects.
Effects of a 2 week course of tDCS on cortical/inhibition balance | Approximately 2 weeks after baseline
  TMS using single and paired pulse paradigms, such as LICI and SICI, will be repeated after completion of the 2 week course of tDCS.
Change in clinical symptoms of agitation as assessed by the Clinical Global Impression of Change (CGIC) | Approximately 2 and 4 weeks after baseline
  The clinical symptoms will be assessed at baseline, after completion of the tDCS intervention and at follow up 2 weeks after last tDCS session. CGIC scores range from 0-7, higher scores indicating worsening compared to baseline.
Change in clinical symptoms of agitation as assessed by the Neuropsychiatric Inventory (NPI) agitation/aggression subscale score | Approximately 2 and 4 weeks after baseline
  The clinical symptoms will be assessed at baseline, after completion of the tDCS intervention and at follow up 2 weeks after last tDCS session. NPI frequency of symptoms are rated on a scale of 0 - 4 (Higher scores indicate symptoms occur more frequently). Severity / intensity of symptoms are rated on a scale of 0 to 3 (Higher scores indicate greater severity of symptoms). Caregiver distress is rated on a scale of 0 to 5 (Higher scores indicate increased caregiver distress).
Change in clinical symptoms of agitation as assessed by the Cohen Mansfield Agitation Inventory scores (CMAI) | Approximately 2 and 4 weeks after baseline
  The clinical symptoms will be assessed at baseline, after completion of the tDCS intervention and at follow up 2 weeks after last tDCS session. CMAI-frequency score ranges between 29 to 203 and CMAI-disruptiveness ranges from 29 to 145 for each category. Higher scores indicate worsening of symptoms.
Assess brain structure using Magnetic Resonance Imaging (MRI) | Baseline
  Brain structure (e.g. cortical atrophy and white matter integrity) will be compared between the 3 groups (AD, AD+agitation and healthy comparators).
Assess resting state connectivity using Functional Magnetic Resonance Imaging (fMRI) | Baseline
  Resting state connectivity using Brain Oxygen Level Dependent (BOLD) signal will be compared between the 3 groups (AD, AD+agitation and healthy comparators).
Assess GABA and glutamate levels using Magnetic Resonance Spectroscopy (MRS) | Baseline
  GABA and glutamate concentrations will be measured in the left DLPFC and compared between the 3 groups (AD, AD+agitation and healthy comparators).

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kumar, MD, FRCPC, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada